CLINICAL TRIAL: NCT05023174
Title: A Randomized Pilot Trial of Platelet Rich Plasma Use in Hiatal Hernia Repair
Brief Title: Platelet Rich Plasma in Hiatal Hernia Repair
Acronym: PPR-HHR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, John Lipham, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APP-20-05449
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hiatal Hernia Large; Reflux, Gastroesophageal
Keywords: platelet rich plasma; hiatal hernia; fundoplication; mesh
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into a treatment arm and a control arm
Who Masked: Participant, Outcomes Assessor
Masking Description: The research personnel will be aware of whether the patient is in the treatment or control arm. The patient will be blinded from this knowledge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP (Experimental): Patients in this treatment arm will have PRP injected into the crura of the diaphragm and coating the mesh placed during the hiatal hernia repair.
  Interventions: Procedure: Hiatal Hernia Repair with Platelet Rich Plasma
- No PRP (Active Comparator): Patients in this arm will undergo an identical surgical procedure, however will not have the addition of PRP injected into the cura of the diaphragm or onto the mesh placed during the hiatal hernia repair.
  Interventions: Procedure: Hiatal Hernia Repair without Platelet Rich Plasma

INTERVENTIONS:
Procedure: Hiatal Hernia Repair with Platelet Rich Plasma — Platelet rich plasma will be injected into the crura of the diaphragm and coating the mesh placed during surgery.
  Arms: PRP
Procedure: Hiatal Hernia Repair without Platelet Rich Plasma — Surgery will be performed without the addition of platelet rich plasma injection
  Arms: No PRP

SUMMARY:
Rationale: Gastroesophageal reflux disease (GERD) is a common disease caused by a dysfunctional lower esophageal sphincter and an abnormal esophageal hiatus or hiatal hernia. Approximately 30% of large hiatal hernias will recur after surgery, in part due to weak connective tissue at the hiatus. Platelet rich plasma (PRP) is a promising autologous therapy that may address this shortcoming by substantially enhancing wound healing of the hiatus after repair.

Intervention: PRP will be applied to mesh used in hiatal hernia repair.

Objectives: The objective of this study is to determine the efficacy of PRP in hiatal hernia compared to traditional hernia repair without PRP.

Study population: 150 patients 18 years and older with large (>5cm) paraesophageal hernias.

Study methodology and study arms: a 1:1 allocation ration will be used to randomly assign 75 patients to the experimental arm (PRP with mesh) and 75 patients to the control arm (mesh only).

Study outcomes: The primary outcome will be 1-year postoperative hernia recurrence based on video esophagram and/or upper endoscopy. The secondary outcome will be GERD-Health Related Quality of Life (GERD-HRQL) scores and dysphagia scores at 6 and 12 months.

Follow-up: Patients who undergo fundoplication and hiatal hernia repair with mesh are seen in clinic for follow-up at two weeks, six weeks, six months, one year, and annually thereafter. Video esophagram or upper endoscopy will be performed at 1 year after surgery to assess the primary outcome. The investigators secondary outcome of reduction in GERD-HRQL score will be determined by a difference in the GERD-HRQL score from the preoperative score to the postoperative scores taken at 6 months and 1 year. The investigators secondary outcome of dysphagia will be determined by EAT-10 scores taken at 6 months and 1 year.

Statistics/Analysis: Descriptive statistics will be used. Intention to treat and per protocol analyses will be performed. Frequentist and Bayesian statistical analyses will be used to determine statistically and clinically important outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Documented hiatal hernia > 5cm on preoperative video esophagram or upper endoscopy

Exclusion Criteria:

* Non-English speaking patients
* Prior antireflux surgery
* Platelet count less than 100,000
* History of platelet dysfunction
* Antiplatelet therapy up to ten days prior to surgery
* Corticosteroids use up to one month before surgery
* Diabetes
* Active malignancy or treatment for cancer within the last year
* Pregnancy or active breastfeeding
* Active smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence on postoperative upper endoscopy or video esophagram | one year
  A hernia of 2 cm or greater on postoperative endoscopy or video esophagram will indicate a recurrence of hiatal hernia

SECONDARY OUTCOMES:
Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) survey score | 6 and 12 months
  GERD quality of life survey responses range from 0-50. A higher score indicated poorer quality of life related to GERD symptoms.
Proton Pump Inhibitor Use | 6 and 12 months
  Reduction in the use of acid-suppressing medications

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Keck Hospital of USC, Los Angeles, California
  - Hoag Hospital, Newport Beach, California